CLINICAL TRIAL: NCT01598792
Title: REALISTIC: A Phase I, Dose Escalation Trial Of Recombinant Listeria Monocytogenes (Lm)-Based Vaccine Encoding Human Papilloma Virus Genotype 16 Target Antigens (ADXS11-001) In Patients With HPV-16 +ve Oropharyngeal Carcinoma
Brief Title: Safety Study of Recombinant Listeria Monocytogenes(Lm)Based Vaccine Virus Vaccine to Treat Oropharyngeal Cancer
Acronym: REALISTIC:
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Patient 2 suffered DLT post-vaccination. The vaccine manufacturers withdrew support for the study on commercial grounds.
Sponsor: University of Liverpool (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government); Cancer Research UK (Other); Advaxis, Inc. (Industry); Recipharm AB (Unknown)
Responsible Party: Principal Investigator, Prof. Terry Jones, Professor of Head and Neck Surgery, University of Liverpool
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISRCTN47069182; 2010-019916-20 (EudraCT Number)
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: HPV-16 +ve Oropharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: ADXS11-001 — Escalating doses will be administered: 3.3 x 10e8,1 x 10e9 and 3.3 x 10e9 cfu to patient in 3 different groups. Dose-escalation will only occur if fewer than two patients in each group of six experience Dose Limiting Toxicity (DLT).

SUMMARY:
It is the investigators intention to investigate whether a specially designed vaccine, based on a genetically modified strain of the bacterium Listeria monocytogenes and called ADXS11-001 is safe to use and is able to boost the immune system of patients presenting with Human Papilloma Virus (HPV) associated oropharyngeal cancer (OPSCC). It is hoped that the vaccine will boost the immune system so that immune cells with cell killing properties are able to attack any cancer cells remaining after the patients have been treated. However, the vaccine is so novel the investigators are not sure whether it is able to do this and before they can answer that question in a larger group of patients they need to make sure that the vaccine is safe to use and has some effect on the immune system in the patients for whom they intend its ultimate use. In a previous study, patients with incurable cervix cancer which is caused by the same virus, were vaccinated with ADXS11-001. Although all patients vaccinated experienced flu-like symptoms, patients tolerated the vaccine well with no patient suffering long term adverse effects of vaccination. However, because the patients and cancer type was so different in this earlier study, the investigators need to test whether ADXS11-001 is also safe in patients with HPV associated OPSCC. That said, the earlier study guided the dosing schedule for the current study and patients entering the REALISTIC trial will receive lower doses than those administered to patients in the earlier cervix cancer study. It is hoped that by doing this, patients will experience fewer side effects of vaccination without reducing the chances of stimulating the immune system.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HPV-16 +ve, p16 +ve OPSCC.
* Patients in remission from disease, i.e. complete response (CR) or unconfirmed complete response (CRu) in the case of non-surgical treatment or complete macroscopic resection of tumour and associated cervical lymph nodes in patients undergoing surgery.
* Completion of standard therapy for malignancy at least 6 weeks before trial entry.
* A positive result following anergy testing.
* Written informed consent and the ability of the patient to co-operate with treatment and follow up must be ensured and documented.
* Age greater than 18 years.
* World Health Organisation (WHO) performance status of 0 or 1.
* Life expectancy of at least 12 months.
* Haematological and biochemical indices (these measurements must be performed within 8 days prior to the patient going on study):
* Haematological:

Haemoglobin (Hb) > 10.0 g/dl Neutrophils ≥ 1.5 x 10e9/L Platelets (Plts) ≥ 100 x 10e9/L

* Baseline liver function tests:

Serum bilirubin ≤ 1.5 x upper normal limit Serum alkaline phosphatase, alanine amino-transferase (ALT) and/or aspartate amino-transferase (AST) < 1.5 x ULN.

* Baseline renal function test:

Calculated creatinine clearance > 50ml/min (uncorrected value) or isotope clearance measurement > 50ml/min.

* Female patients of child-bearing potential are eligible, provided they have a negative serum pregnancy test prior to enrolment and agree to use appropriate medically approved contraception during the study up to six months after the last vaccination Male patients must agree to use appropriate medically approved contraception during the study up to six months after the last vaccination.

Exclusion Criteria:

* Receiving, or having received, chemotherapy or radiotherapy within 6 weeks of trial entry.
* Having undergone surgery +/- PORT within 6 weeks of trial therapy
* A negative result following anergy testing.
* Known chronic active infection with Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV).
* Current active autoimmune disease.
* Current active skin diseases requiring therapy (psoriasis, eczema etc).
* Ongoing active infection.
* History of anaphylaxis or severe allergy to vaccination.
* Previous myeloablative therapy followed by an autologous or allogeneic haematopoietic stem cell transplant.
* Patients who have had a splenectomy or splenic irradiation, or with known splenic dysfunction.
* Receiving current immunosuppressive medication, including corticosteroids within 4 weeks of the first dose.
* Pregnant and lactating women.
* Ongoing toxic manifestations of previous treatment.
* Major thoracic and/or abdominal surgery in the preceding four weeks from which the patient has not yet recovered.
* Patients with any other condition which in the Investigator"s opinion would not make the patient a good candidate for the clinical trial.
* Concurrent congestive heart failure or prior history of class III/ IV cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety | 12 months
  Occurrence of drug-related grade 3 or 4 systemic or local adverse events (defined using the NCI Common Criteria Adverse Events (CTCAE) Version 4.03

SECONDARY OUTCOMES:
Translational | 24 Months
  Demonstration by ELISPOT assay of the frequency of IFN-γ secreting lymphocytes recognising MHC class I and II-restricted epitopes within HPV-16 E& protein in peripheral blood at sequential time-points before, during and up to ten months after vaccination course. This protocol has been used by our group to demonstrate vaccine induced T cell responses in a previous HPV vaccine trial.

CONTACTS AND LOCATIONS:
Overall Officials: Terence Jones, BSc,FRCS,MD, Principal Investigator — University of Liverpool
Locations (4):
- United Kingdom (4):
  - Velindre NHS Trust, Cardiff
  - The Royal Liverpool and Broadgreen University Hospitals NHS Foundation Trust, Liverpool
  - Aintree University NHS Foundation Trust, Liverpool
  - The Royal Marsden NHS Foundation Trust, London

REFERENCES:
- See also: Cancer Research UK — http://www.cancerresearchuk.org/
- See also: Liverpool Cancer Trials Unit — http://www.lctu.org.uk